CLINICAL TRIAL: NCT05003960
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Autism
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for Autism
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-8-ATG-8-02
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Autism
Keywords: Autism; stem cell treatment
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): One intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Autism

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Autism. Patients with Autism will receive a single intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells. The total dose for the infusion will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety
* Previous organ transplant
* Seizure disorder
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: Autism Treatment Evaluation Checklist (ATEC) | Four year follow-up
  ATEC is a questionnaire to measure changes in severity in response to treatment. It will be completed for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (3):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Greece (2):
  - Athens Beverly Hills Medical Group, Glyfada, Athens
  - Mediterraneo Hospital Ilias 8-12, Glyfada, Athens

REFERENCES:
- [Background] Mahapatra S, Vyshedsky D, Martinez S, Kannel B, Braverman J, Edelson SM, Vyshedskiy A. Autism Treatment Evaluation Checklist (ATEC) Norms: A "Growth Chart" for ATEC Score Changes as a Function of Age. Children (Basel). 2018 Feb 16;5(2):25. doi: 10.3390/children5020025. PMID 29462954
- [Background] Lv YT, Zhang Y, Liu M, Qiuwaxi JN, Ashwood P, Cho SC, Huan Y, Ge RC, Chen XW, Wang ZJ, Kim BJ, Hu X. Transplantation of human cord blood mononuclear cells and umbilical cord-derived mesenchymal stem cells in autism. J Transl Med. 2013 Aug 27;11:196. doi: 10.1186/1479-5876-11-196. PMID 23978163
- [Background] Riordan NH, Hincapie ML, Morales I, Fernandez G, Allen N, Leu C, Madrigal M, Paz Rodriguez J, Novarro N. Allogeneic Human Umbilical Cord Mesenchymal Stem Cells for the Treatment of Autism Spectrum Disorder in Children: Safety Profile and Effect on Cytokine Levels. Stem Cells Transl Med. 2019 Oct;8(10):1008-1016. doi: 10.1002/sctm.19-0010. Epub 2019 Jun 11. PMID 31187597 (Retraction: PMID 34847283 Stem Cells Transl Med. 2021 Dec;10(12):1717)